CLINICAL TRIAL: NCT02082717
Title: The Impact of 4% Sodium Bicarbonate Additive During Potassium Chloride Replacement on Pain and Incidence of Phlebitis for Adult Patients in a Medical Surgical Unit: A Randomized Double Blinded Controlled Study
Brief Title: The Impact of Neut During Potassium Chloride Replacement on Pain and Incidence of Phlebitis
Acronym: Neut-WKBH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to medical supplies shortages due to the 2017 hurricane season.
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB # 13-060
Record Dates: First submitted 2014-02-24; First posted 2014-03-10 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hypokalemia
MeSH Terms: conditions — Hypokalemia | interventions — Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neut (4%sodium bicarbonate additive) (Experimental): 4% sodium bicarbonate additive during intravenous potassium chloride replacement.
  Interventions: Drug: potassium chloride replacement; Drug: Experimental - 4% Sodium Bicarbonate
- Control (Active Comparator): standard of practice potassium chloride replacement (with no additive)
  Interventions: Drug: potassium chloride replacement

INTERVENTIONS:
Drug: potassium chloride replacement
Drug: Experimental - 4% Sodium Bicarbonate
  Arms: Neut (4%sodium bicarbonate additive)

SUMMARY:
The purpose of this study is to examine the impact of 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy for adult patients in a Medical/Surgical unit. Using a randomized controlled double blinded experimental study design, patients who are 21 years or older are alert, awake, and oriented at the time of enrollment and have been ordered peripheral intravenous potassium chloride replacement will be recruited from one Medical/Surgical during the first 24-48 hours of their admission.

DETAILED DESCRIPTION:
The specific aim of the study is:

Aim 1: To compare patient outcomes (phlebitis, pain at peripheral IV insertion site, frequency of changing IV access, and time for administration) between the experimental (4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy) and control (standard of practice of no 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy) groups.

Aim 2: To compare number and type of nursing interventions done during peripheral intravenous potassium chloride replacement therapy between the experimental (4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy) and control (standard of practice of no 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy) groups.

Aim 3: To compare attrition rates and reasons between the experimental (4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy) and control (standard of practice of no 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy) groups.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the medical/surgical unit within the last 24 to 48 hours
* awake, alert, and oriented times three
* 21 years old and greater
* receiving first peripheral intravenous potassium chloride replacement therapy as ordered by physician or ARNP as part of care and regardless of research
* potassium level of 3.5 mmol/L or less.

Exclusion Criteria:

* patients who have been in the medical/surgical unit more than 48 hours.
* altered mental status defined as not being awake, alert, and oriented times three
* patients who already received intravenous potassium chloride replacement during the current admission and with the current IV access
* patients receiving intravenous potassium replacement therapy through a central line
* patients that are not ordered potassium replacement by physician or ARNP as part of their care while hospitalized.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mavel Arinal, RN, Principal Investigator — BHSF
Locations (1):
- West Kendall Baptist Hospital, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Neut (4%Sodium Bicarbonate Additive): 4% sodium bicarbonate additive during intravenous potassium chloride replacement.
  potassium chloride replacement
  Experimental - 4% Sodium Bicarbonate
- Control: standard of practice potassium chloride replacement (with no additive)
  potassium chloride replacement
Period: Overall Study
Arm/Group | Neut (4%Sodium Bicarbonate Additive) | Control
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neut (4%Sodium Bicarbonate Additive) | Control | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 3 | 5 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Indicated Findings
Description: outcomes - phlebitis, pain at peripheral intravenous insertion site, frequency of changing IV access, and time for administration.
  experimental - 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy.
  control - standard of practice of no 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy.
Time Frame: Up to 4 hours
Population: Due to the small number of participants enrolled, the statistical power would be too low for any significant findings.
Measure: Count of Participants; unit: Participants
Arm/Group | Neut (4%Sodium Bicarbonate Additive) | Control
Number analyzed (Participants) | 8 | 9
Participants
  Pain at 15 min. at IV site | 0 | 1
  Pain at 1 hour at IV site: number analyzed (Participants) | 7 | 9
  Pain at 1 hour at IV site | 1 | 0
  Pain at 2 hours at IV site: number analyzed (Participants) | 4 | 5
  Pain at 2 hours at IV site | 0 | 2
  Pain at 3 hours at IV site: number analyzed (Participants) | 2 | 4
  Pain at 3 hours at IV site | 1 | 2
  Pain at 4 hours at IV site: number analyzed (Participants) | 2 | 4
  Pain at 4 hours at IV site | 0 | 0
  Pain at completion: number analyzed (Participants) | 3 | 7
  Pain at completion | 0 | 0
  Phlebitis (Erythema and Swelling at IV site) at 15 mins. | 0 | 1
  Phlebitis (Erythema and Swelling at IV site) at 1 hour: number analyzed (Participants) | 7 | 8
  Phlebitis (Erythema and Swelling at IV site) at 1 hour | 0 | 0
  Phlebitis (Erythema and Swelling at IV site) at 2 hours: number analyzed (Participants) | 4 | 5
  Phlebitis (Erythema and Swelling at IV site) at 2 hours | 0 | 0
  Phlebitis (Erythema and Swelling at IV site) at 3 hours: number analyzed (Participants) | 2 | 4
  Phlebitis (Erythema and Swelling at IV site) at 3 hours | 0 | 0
  Phlebitis (Erythema and Swelling at IV site) at 4 hours: number analyzed (Participants) | 2 | 4
  Phlebitis (Erythema and Swelling at IV site) at 4 hours | 0 | 0
  Slight pain and redness at IV site at 15 min | 1 | 3
  Slight pain and redness at IV site at 1 hour: number analyzed (Participants) | 7 | 8
  Slight pain and redness at IV site at 1 hour | 3 | 2
  Slight pain and redness at IV site at 2 hours: number analyzed (Participants) | 4 | 5
  Slight pain and redness at IV site at 2 hours | 0 | 2
  Slight pain and redness at IV site at 3 hours: number analyzed (Participants) | 2 | 4
  Slight pain and redness at IV site at 3 hours | 0 | 1
  Slight pain and redness at IV site at 4 hours: number analyzed (Participants) | 2 | 4
  Slight pain and redness at IV site at 4 hours | 1 | 0
  Slight pain and redness at IV site at completion: number analyzed (Participants) | 3 | 7
  Slight pain and redness at IV site at completion | 1 | 0

2. Secondary Outcome: Number of Participants Nursing Interventions
Description: experimental - 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy
  control - standard of practice of no 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy
Time Frame: Up to 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Neut (4%Sodium Bicarbonate Additive): 4% sodium bicarbonate additive during intravenous potassium chloride replacement.
  potassium chloride replacement
  Experimental - 4% Sodium Bicarbonate
  3 participants out of 8 analyzed had pain medication during randomization.
- Control: standard of practice potassium chloride replacement (with no additive)
  potassium chloride replacement
  O participants out of 9 had no interventions
Arm/Group | Neut (4%Sodium Bicarbonate Additive) | Control
Number analyzed (Participants) | 8 | 9
Participants
  Nursing Intervention - Pain medication | 3 | 0
  No nursing intervention | 5 | 9

3. Secondary Outcome: Attrition Rates
Description: experimental - 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy.
  control - standard of practice of no 4% sodium bicarbonate additive during peripheral intravenous potassium chloride replacement therapy
Time Frame: Up to 4 hours
Measure: Count of Participants; unit: Participants
Groups:
- Neut (4%Sodium Bicarbonate Additive): 4% sodium bicarbonate additive during intravenous potassium chloride replacement.
  potassium chloride replacement
  Experimental - 4% Sodium Bicarbonate
  Zero attrition rate
- Control: standard of practice potassium chloride replacement (with no additive)
  potassium chloride replacement
  Zero attrition rate
Arm/Group | Neut (4%Sodium Bicarbonate Additive) | Control
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 4 hours
Arm/Group | Neut (4%Sodium Bicarbonate Additive) | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT02082717/Prot_SAP_000.pdf